CLINICAL TRIAL: NCT00386854
Title: Metabolic Study of Concentric and Eccentric Muscle Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vorarlberg Institute for Vascular Investigation and Treatment (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: K01-2003-1
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2006-10-12 (Estimated); Status verified 2006-10

CONDITIONS: Lipid Metabolism; Insulin Resistance; Inflammation
Keywords: exercise; lipid metabolism; lipoproteins; insulin resistance; inflammation
MeSH Terms: conditions — Insulin Resistance; Inflammation; Motor Activity | interventions — Physical Conditioning, Human

INTERVENTIONS:
Behavioral: physical training

SUMMARY:
The purpose of this study is to evaluate the metabolic and anti-inflammatory effects of eccentric endurance exercise and to compare them with those of concentric exercise in healthy sedentary individuals.

DETAILED DESCRIPTION:
Physical exercise decreases the risk of obesity, diabetes mellitus, and cardiovascular disease. Skeletal muscle can be exercised by two ways: Concentric contraction is defined as active shortening of muscles, e.g. by stepping upwards, whereas eccentric muscle contraction is defined as active resistance to stretching, e.g. by stepping downwards. Although the effects of exercise (i.e. the combination of concentric and eccentric muscle contraction) on metabolic parameters have been extensively investigated, there are no data on the specific metabolic effects of concentric versus those of eccentric muscle work in humans.

Comparison(s): Metabolic and anti-inflammatory effects of eccentric endurance exercise (i.e. stepping upwards), compared to metabolic and anti-inflammatory effects of concentric exercise (i.e. stepping downwards).

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women
* age over 30 years

Exclusion Criteria:

* previous systematic endurance training (≥3 times per week ≥30 min)
* body mass index >30 kg/m2
* heavy smoking (>20 cigarettes per day)
* regular alcohol consumption >60g per day
* established musculoskeletal disease
* history of cardiovascular disease
* diabetes mellitus
* unwillingness to stay in the area for the whole study period

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-04; Study Completion 2003-08

PRIMARY OUTCOMES:
Metabolic and anti-inflammatory effects induced by eccentric muscle exercise.

SECONDARY OUTCOMES:
Metabolic and anti-inflammatory effects induced by concentric muscle exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Drexel, MD, Principal Investigator — Vorarlberg Institut of Vascular Investigation and Treatment, Academic Teaching Hospital, Austria
Locations (1):
- Vorarlberg Institute of Vascular Investigation and Treatment, Feldkirch, Vorarlberg, Austria

REFERENCES:
- [Derived] Drexel H, Mader A, Saely CH, Tautermann G, Dopheide JF, Vonbank A. Downhill hiking improves low-grade inflammation, triglycerides, body weight and glucose tolerance. Sci Rep. 2021 Jul 15;11(1):14503. doi: 10.1038/s41598-021-93879-1. PMID 34267272